CLINICAL TRIAL: NCT01956318
Title: Crenobalneotherapy in the Treatment of Chronic Venous Insufficiency. A Randomized Clinical Trial.
Brief Title: Crenobalneotherapy in the Treatment of Chronic Venous Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre de Recherche Rhumatologique et Thermal (Other)
Responsible Party: Principal Investigator, FORESTIER Romain, President of the research center, Centre de Recherche Rhumatologique et Thermal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Thermes2010
Record Dates: First submitted 2013-09-29; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Balneology
Keywords: Chronic venous insufficiency; Varicose vein; Crenobalneotherapy; Balneotherapy; Spa therapy
MeSH Terms: conditions — Varicose Veins | interventions — Balneology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crenobalneotherapy (Experimental): 18 days of balneotherapy session in 3 weeks. Patients are also delivered a booklet with advice on lifestyle.
  Interventions: Behavioral: Crenobalneotherapy
- control group (No Intervention): patients are allowed to continue their usual drugs, compression therapy and are delivered a booklet with advice on lifestyle.

INTERVENTIONS:
Behavioral: Crenobalneotherapy — 18 days of balneotherapy session in 3 weeks. Each day, the treatment associates 4 techniques: Kneipp Therapy, walking pool, underwater massage, bath tub and finishing with 20 minutes of rest in the Trendelendburg position. Kneipp Therapy is an alternating warm (28°C) and cold (14°C) shower on the legs during 10 minutes. Walking pool is a 60 cm deep pool at 23°C with underwater shower where patients are walking without stopping during 10 minutes. Underwater massage is realized by a senior physiotherapist. It starts at the feet and gradually rises to the thighs during 10 minutes. Bath tub is underwater shower at 30°C. It also starts at the feet and gradually rises to the thighs during 20 minutes. The interventions are standardized by timers. Adherence to each technique is supervised before each session in the usual manner for each patient treated in the spa center.
  Other Names: Crenotherapy; Balneotherapy; Spa therapy
  Arms: Crenobalneotherapy

SUMMARY:
At 3 months, crenobalneotherapy session is superior to waiting list for patients with chronic venous insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 80 years with chronic venous insufficiency regardless of etiology stages 3 or 4 according to the CEAP classification (Clinical severity, Etiology or cause, Anatomy, Pathophysiology)
* Patients available to participate in a 3 weeks session in the spa center and to be followed for 6 months

Exclusion Criteria:

* pregnant women,
* contra-indication for the spa treatment (chronic infectious diseases, cancer, heart failure, serious liver or kidney disease, open leg ulcer, psychiatric disorders, immune deficiency, phlebitis, erysipelas or history of erysipelas);
* surgery in the next three months,
* spa treatment in the previous 6 months,
* professional involvement with a spa resort

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
number of patient with 20% improvement of CIVIC scale at 3 months | 3 months
  Primary outcome is the number of patient with 20% improvement in quality of life (CIVIC scale) at 3 months

SECONDARY OUTCOMES:
CIVIC | 1 month
  Chronic Venous Insufficiency Questionnaire (CIVIQ 2) 20% improvement. disease-specific QOL score for patients with chronic venous disease. The total score is derived from 20 questions (items) that represent four QOL dimensions (of 3-9 items each): bodily pain, physical, social and psychological functioning. The possible scores for each item are as follows: 1, negative; 2, weak; 3, moderate; 4, strong; 5, severe. The total scores can therefore vary from 20 (no symptoms) to 100 (worse possible condition).
civic | 1 & 3 months
  evolution of civic scale
Rutherford severity score | 1 & 3 months
  clinical evaluation of severity taking into account 10 attributes: pain, varicose veins, venous edema, skin pigmentation, and adherence to compressive therapy, inflammation, induration, number, size and duration of active ulcer. Each attribute is scored 0 (minimum) to 2 (maximum).
PASS | 1 & 3 months
  PASS is measured by asking the patient if he/she feels he/she is in an acceptable clinical condition in terms of its venous insufficiency. We measure the number of patients with PASS
opinion of patient and practitionner | 1 & 3 months
  Opinion of patient and practitioner is determined on a 5 point Lickert scale (very aggravated, aggravated, unchanged, improved and very improved)
associated treatment | 1 & 3 months
  Drug consumption is estimated on the last 3 days prior to the evaluation. Surgery, hospitalization for venous insufficiency and adherence to compression therapy
side effects | week 1 & 3. 1 & 3 months
  side effects are collected by therapists and assessor. we collected the number of patients with side effects and the type of side effect

REFERENCES:
- [Derived] Forestier RJ, Briancon G, Francon A, Erol FB, Mollard JM. Balneohydrotherapy in the treatment of chronic venous insufficiency. Vasa. 2014 Sep;43(5):365-71. doi: 10.1024/0301-1526/a000374. PMID 25147013